CLINICAL TRIAL: NCT07319247
Title: The Effect of High-frequency Laser Therapy and Pelvic Floor Muscle Training in Women With Stress Urinary Incontinence: A Plasebo Randomized Controlled Trial
Brief Title: Laser Therapy and Pelvic Floor Muscle Training for Stress Urinary Incontinence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, hanife dogan, Physıcal Therapy and Rehabilitation, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hlaser
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence (UI); Laser Therapy; Stress Urinary Incontinence (SUI); Pelvic Floor Muscle Exercise
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PFME Group (Active Comparator): In this training, patients are taught pelvic floor exercises, which involve slow and fast muscle contractions that train both Type 1 and Type 2 muscle fibers, using vaginal palpation. During fast contractions, patients are asked to quickly contract and relax their pelvic floor muscles. The image of "turning the faucet off and on" is used to help patients better understand this exercise. During slow contractions, patients are asked to slowly tighten their pelvic floor muscles, hold them for 10 seconds, and then slowly relax them. One set of pelvic floor muscle exercises consists of 10 fast contractions and 10 slow contractions. According to this program, pelvic floor exercises are performed in weeks 1-2, 2 sets in weeks 3-4, 4 sets in weeks 5-6, 8 sets in weeks 7-8, and 10 sets in weeks 8-12. Assessments will be conducted twice, baseline and post treatment (at 10 week).
  Interventions: Behavioral: PFMT Group
- PFME+Laser (Active Comparator): PFMT, patients are taught pelvic floor exercises, which involve slow and fast muscle contractions that train both Type 1 and Type 2 muscle fibers, using vaginal palpation. During fast contractions, patients are asked to quickly contract and relax their pelvic floor muscles. The image of "turning the faucet off and on" is used to help patients better understand this exercise. During slow contractions, patients are asked to slowly tighten their pelvic floor muscles, hold them for 10 seconds, and then slowly relax them. One set of pelvic floor muscle exercises consists of 10 fast contractions and 10 slow contractions. Assessments will be conducted twice, baseline and post treatment (at 10 weeks). Laser was also applied to this group. Laser application is applied to 6 points in the perineal area. Continue and biostimulatory mode, intensity 6W, energy density 120J/cm2. Application time is 2 minutes for each point, and a total of 6 sessions are applied 3 time.
  Interventions: Behavioral: PFME+Laser Therapy
- Plasebo Laser (Placebo Comparator): This group will only receive placebo laser treatment. The sound will be turned up as if the laser is being applied, but no warning will be given. The laser device will be aimed at 6 points in the perineal area without being plugged in. Assessments will be conducted twice, baseline and post treatment (at 10 weeks).
  Interventions: Other: Plasebo Laser

INTERVENTIONS:
Behavioral: PFME+Laser Therapy — PFMT, patients are taught pelvic floor exercises, which involve slow and fast muscle contractions that train both Type 1 and Type 2 muscle fibers, using vaginal palpation. During fast contractions, patients are asked to quickly contract and relax their pelvic floor muscles. The image of "turning the faucet off and on" is used to help patients better understand this exercise. During slow contractions, patients are asked to slowly tighten their pelvic floor muscles, hold them for 10 seconds, and then slowly relax them. One set of pelvic floor muscle exercises consists of 10 fast contractions and 10 slow contractions. According to this program, pelvic floor exercises are performed in weeks 1-2, in weeks 3-4, in weeks 5-6, in weeks 8-12, and in weeks 10.
  Laser application is applied to 6 points in the perineal area. Continue and biostimulatory mode, intensity 6W, energy density 120J/cm2. Application time is 2 minutes for each point, and a total of 6 sessions are applied 3 time
  Arms: PFME+Laser
Other: Plasebo Laser — The laser device will be held on 6 points in the perineal area for the same period of time without being plugged in.
  Arms: Plasebo Laser
Behavioral: PFMT Group — In this training, patients are taught pelvic floor exercises, which involve slow and fast muscle contractions that train both Type 1 and Type 2 muscle fibers, using vaginal palpation. During fast contractions, patients are asked to quickly contract and relax their pelvic floor muscles. The image of "turning the faucet off and on" is used to help patients better understand this exercise. During slow contractions, patients are asked to slowly tighten their pelvic floor muscles, hold them for 10 seconds, and then slowly relax them. One set of pelvic floor muscle exercises consists of 10 fast contractions and 10 slow contractions. According to this program, pelvic floor exercises are performed in weeks 1-2, 2 sets in weeks 3-4, 4 sets in weeks 5-6, 8 sets in weeks 7-8, and 10 sets in weeks 8-12. Assessments will be conducted twice, baseline and post treatment (at 10 week).
  Arms: PFME Group

SUMMARY:
The aim of this study was to investigate the effects of Pelvic Floor Muscle Training (PFMT) in addition to high-intensity laser therapy (HILT) on pelvic floor dysfunction, sexual dysfunction, and quality of life in women with stress urinary incontinence. Women with SUI will be randomly assigned to PFMT (Group I), Laser + PFMT (Group II), and placebo laser (Group III). PFMT will be administered twice weekly for 10 weeks under the supervision of a physiotherapist. PFMT will be administered with biofeedback. HFMT will be applied to six points in the perineal region (2 minutes per point). The intensity will be 6W, the energy density will be 120J/cm2, and three sessions will be administered weekly for a total of six sessions. Women included in the study will be evaluated twice, at the beginning and at the end of the treatment, with the Incontinence Quality of Life Scale (I-QOL), Incontinence Severity Index (ISI), Female Sexual Function Scale-(FSFI), and Global Pelvic Floor Impact Questionnaire (GPTRA).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65,
* Women who are volunteers and committed to work,
* Women diagnosed with stress urinary incontinence,

Exclusion Criteria:

* Pregnancy,
* Previous surgery in the treatment area within 12 months,
* Active genital infection,
* Presence of malignancy,
* Systemic steroid use in the last 3 months,
* Use of vaginal lubricant within the last 7 days,
* Recurrent urinary tract or genital herpes,
* POP-Q score 3 or higher

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence severity | baseline, post treatment (at 10 week)
  The Incontinence Severity Index (ISI): This is a two-question questionnaire that helps calculate the severity of urinary incontinence in patients. It categorizes incontinence severity into three groups: mild, moderate, and severe. It is a useful method for monitoring and assessing incontinence severity.
The impact of urinary incontinence on quality of life | baseline, post treatment (at 10 week)
  The Incontinence Quality of Life Scale (I-QOL) will be used to determine the impact of urinary incontinence on quality of life in women. It consists of questions under three headings: behavioral, psychological, and social impact. The questions will be asked of the participants and recorded.
pelvic floor dysfuntion severity | baseline, post treatment (at 10 week)
  The Global Pelvic Floor Impact Questionnaire (GPTRA): This questionnaire consists of nine questions addressing pelvic floor dysfunction. A higher total score indicates a greater degree of symptoms. Participants were asked questions and recorded.

SECONDARY OUTCOMES:
Sexually Dysfunction | baseline, post treatment (at 10 week)
  The Female Sexual Function Index (FSFI): It consists of nineteen separate questions. It has six subscales: desire, arousal, lubrication, orgasm, general satisfaction, and pain. Questions 3-14 and 15-19 are scored on a 6-point Likert-type scale (0-5), while the remaining questions are scored on a 5-point Likert-type scale (1-5). The scale, which can be applied to those who have had sexual intercourse within the last month, is scored negatively, with higher scores interpreted as indicating no or low sexual dysfunction. The highest possible score is 36.0, and the lowest is 2.0. The cut-off score is 26.55.
  Scores of 26.55 and below are considered to indicate sexual dysfunction.
pelvic floor muscle function | baseline, post treatment (at 10 week)
  Pelvic floor muscle function will be assessed with EMG biofeedback.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy Hospital, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No